CLINICAL TRIAL: NCT06913504
Title: Comparison Of Blue Light Filter Feature and Blue Blocking Lenses in Digital Device Users With Dry Eye Patients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MSRSW/Batch-Fall23/804
Record Dates: First submitted 2025-03-29; First posted 2025-04-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-03

CONDITIONS: Dry Eye Syndromes
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Blue cut filter (Experimental)
  Interventions: Diagnostic Test: Blue cut filter
- blue cut glasses (Experimental)
  Interventions: Diagnostic Test: blue cut glasses

INTERVENTIONS:
Diagnostic Test: Blue cut filter — Group 1 will be prescribe with blue cut filter feature
  Arms: Blue cut filter
Diagnostic Test: blue cut glasses — Group 2 will be prescribed with blue cut glasses
  Arms: blue cut glasses

SUMMARY:
Comparing Blue Light Filter feature and Blue Blocking Lenses for Dry Eye Patients Prolonged screen time can exacerbate dry eye symptoms.

DETAILED DESCRIPTION:
Two solutions, blue light filter software and blue blocking lenses, aim to reduce eye strain. Blue light filter software adjusts screen color temperatures, reducing blue light emission. Blue blocking lenses provide a physical barrier, blocking blue light from reaching the eyes.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 12-34
* Spend at least 4 hours per day on digital devices.
* Experience dry eye symptoms.
* Willing to participate in the study and provide informed consent.

Exclusion Criteria:

* Pre-existing eye conditions (e.g., cataracts, glaucoma).
* Wear contact lenses.
* Have undergone eye surgery.
* Are pregnant or breastfeeding.

Ages: 12 Years to 34 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 54 (Actual)
Dates: Start 2025-03-20 (Actual); Primary Completion 2025-06-20 (Estimated); Study Completion 2026-02-20 (Estimated)

PRIMARY OUTCOMES:
The Ocular Surface Disease Index (OSDI) | 12 Months
  The Ocular Surface Disease Index (OSDI) is a 12-question questionnaire used to assess the severity of dry eye symptoms and their impact on vision-related function, scored on a scale of 0 to 100, with higher scores indicating greater disability

CONTACTS AND LOCATIONS:
Locations (1):
- Khursheed baigam eye hospital raiwind road manga mandi, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No